CLINICAL TRIAL: NCT00794196
Title: Impact of the Pharmaceutical Care Program for Pharmacological Treatment of Depression in Primary Care on the Compliance to Antidepressants and Patient Wellbeing
Brief Title: Pharmaceutical Care Program for Pharmacological Treatment of Depression in Primary Care
Acronym: PRODEFAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Carlos III Health Institute (Other Government); Catalan Institute of Health (Other Government); University of Barcelona (Other)
Responsible Party: Principal Investigator, Antoni Serrano Blanco, Antoni Serrano Blanco, Fundació Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FIS PI070546
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-10

CONDITIONS: Depression
Keywords: Medication adherence; Antidepressive agents; Primary care; Pharmaceutical care
MeSH Terms: conditions — Depression; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): The control group will be receiving usual medical and pharmaceutical care.
- Intervention Group (Experimental): Intervention group will be receiving usual medical and pharmaceutical care plus a pharmaceutical support program.
  Interventions: Behavioral: Pharmaceutical care program for antidepressant treatment

INTERVENTIONS:
Behavioral: Pharmaceutical care program for antidepressant treatment — The pharmaceutical care program is a support program for patients starting and maintaining antidepressant treatment.
  Other Names: PRODEFAR group
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to evaluate the impact of pharmaceutical services among patients starting a treatment with antidepressants for a diagnosis of depression. The hypothesis of the study is that pharmacist intervention can improve compliance to antidepressants and patient wellbeing.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of a support program in community pharmacy on the improvement of the compliance to antidepressants and the clinic of typical primary care patients under normal practice circumstances. That implies that the intervention is made by pharmacists without any specific requirement that work in the community pharmacies set up in the area of study and on patients following the usual medical circuit. As well, the cost of the support program is calculated in order to set the effectiveness of the program.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis for depression from a general practitioner
* Beginning a pharmacological antidepressant treatment
* Going to one of the participant community pharmacies

Exclusion Criteria:

* Used antidepressant medication in the past 2 months
* Had an appointment with an specialist in mental disorders in the past 2 months
* History of psychotic or bipolar episodes
* History of drug abuse or dependency
* Cognitive impairment that not allows assessment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Serrano, MD PhD, Principal Investigator — Foundation Sant Joan de Deu
Locations (2):
- Spain (2):
  - Primary Care Center Doctor Bartomeu Fabres Anglada, Gavà, Barcelona
  - Primary Care Center Gavà 1, Gavà, Barcelona

REFERENCES:
- [Derived] Rubio-Valera M, Bosmans J, Fernandez A, Penarrubia-Maria M, March M, Trave P, Bellon JA, Serrano-Blanco A. Cost-effectiveness of a community pharmacist intervention in patients with depression: a randomized controlled trial (PRODEFAR Study). PLoS One. 2013 Aug 12;8(8):e70588. doi: 10.1371/journal.pone.0070588. eCollection 2013. PMID 23950967
- [Derived] Rubio-Valera M, Serrano-Blanco A, Trave P, Penarrubia-Maria MT, Ruiz M, Pujol MM. Community pharmacist intervention in depressed primary care patients (PRODEFAR study): randomized controlled trial protocol. BMC Public Health. 2009 Aug 5;9:284. doi: 10.1186/1471-2458-9-284. PMID 19656386

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: The control group will be receiving usual medical and pharmaceutical care at primary care level. They could be referred to specialized care when necessary (general practitioner's criteria).
Period: Overall Study
Arm/Group | Usual Care | Intervention Group
Started | 92 | 87
Completed | 87 | 64
Not Completed | 5 | 23
Not completed — Lost to Follow-up | 5 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention Group | Total
Number analyzed (Participants) | 92 | 87 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (15.9) | 49.4 (15.1) | 48.9 (15.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 60 | 130
  >=65 years | 22 | 27 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 58 | 135
  Male | 15 | 29 | 44
Region of Enrollment [Number; unit: participants]
  Spain | 92 | 87 | 179

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Antidepressant Medication
Description: Adherence to antidepressant medication was measured through Pharmacy records
Time Frame: At 3 and 6 months
Measure: Number (95% Confidence Interval); unit: percentage of adherence patients
Arm/Group | Intervention Group | Usual Care
Number analyzed (Participants) | 87 | 92
percentage of adherence patients
  3 months | 78.4 [48.0 to 93.5] | 61.9 [26.4 to 88.1]
  6 months | 60.1 [28.4 to 85.11] | 40.2 [12.9 to 75.3]

2. Secondary Outcome: Patient Wellbeing
Description: Patient wellbeing EUROQOL5D scale is used to evaluate health-related quality of life.
  The answers given to EUROQOL5D allow for the description 243 unique health states which can be converted into EQ-5D index anchored at 0 for death and 1 for perfect health.
Time Frame: 0, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Usual Care
Number analyzed (Participants) | 87 | 92
units on a scale
  Baseline | 0.58 [0.50 to 0.65] | 0.66 [0.58 to 0.75]
  3 months | 0.78 [0.70 to 0.86] | 0.79 [0.71 to 0.88]
  6 months | 0.85 [0.76 to 0.93] | 0.80 [0.74 to 0.91]

ADVERSE EVENTS:
Arm/Group | Usual Care | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/87
Other Adverse Events (participants affected / at risk) | 0/92 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No